CLINICAL TRIAL: NCT03701191
Title: Assessment of Postoperative Discomfort Following Inverted Periosteal Pedicle Flap Versus Coronally Advanced Flap With Subepithelial Connective Tissue Graft in Treatment of Gingival Recession Types 1 and 2. A Randomized Clinical Trial.
Brief Title: Using Inverted Periosteal Pedicle Flap in Treatment of Gingival Recession
Acronym: IPPF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marwa El Sayed Abbas Ahmed (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Marwa El Sayed Abbas Ahmed, Assistant Lecturer, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: perio 2:5:1
Record Dates: First submitted 2018-10-07; First posted 2018-10-09 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Gingival Recession
Keywords: gingival recession, periosteum, autogenous graft
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Included participants will be:
  1. Gender: Male and Female
  2. Age: >20 years
  3. Have RT1 and RT2 gingival recession
  Exclusion criteria:
  1. Medically compromised
  2. History of certain medications
  3. Pregnant females
  4. Periapical involvement in selected teeth
  5. History of periodontal surgery involving experimental teeth
  6. If the problem was due to orthodontic treatment
Who Masked: Outcomes Assessor
Masking Description: Two outcome assessors will be chosen: one will be a periodontist but not included within the research; and the other will be a non-periodontist. The outcome assessors will be blinded; they will not be informed by the type of intervention to be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grpup A (Test group) (Experimental): Inverted periosteal pedicle flap will be carried out
  Interventions: Procedure: Inverted periosteal pedicle flap
- Group B (Control group) (Active Comparator): Coronally advanced flap with subepithelial connective tissue graft
  Interventions: Procedure: Inverted periosteal pedicle flap

INTERVENTIONS:
Procedure: Inverted periosteal pedicle flap — The periosteum will be used as an autogenous graft after raising a partial thickness flap in group A

SUMMARY:
Perioteum in the recession defect site will be used as an autogenous graft after raising a flap and the results will be compared with another group which will be treated by the gold standard ( coronally advanced flap with subepithelial connective tissue graft).

DETAILED DESCRIPTION:
Eighteen participants will be recruited.

Included participants will be:

1. Gender: Male and Female
2. Age: >20 years
3. Have RT1 and RT2 gingival recession

Exclusion criteria:

1. Medically compromised
2. History of certain medications
3. Pregnant females
4. Periapical involvement in selected teeth
5. History of periodontal surgery involving experimental teeth
6. If the problem was due to orthodontic treatment

11. Interventions: Participants will be divided into two groups, group A (test group) and group B ( control group).

Pre-surgical phase (including supragingival scaling and root planning) will be carried out to both groups, followed by oral hygiene instructions.

Then, Participants will be explained about each procedure. 7

For group A (test group):

Inverted periosteal pedicle flap will be carried out as follows according to Shetty 2014:

Patients will be explained about the procedure. Non-surgical phase will include supragingival scaling and root planning, followed by oral hygiene instructions.

The surgical procedure will be carried out three weeks after non-surgical phase as follows:

1. Horizontal incisions will be made perpendicular to the adjacent papillae at the level of the cement-enamel junction (CEJ) preserving the gingival margin of the affected teeth.
2. Sulcular incisions on the buccal/facial aspect of the involved teeth.
3. Vertical incisions extending beyond the mucogingival junction will be made at the line angles of the distal most and the mesial most teeth.
4. A partial thickness flap will then be elevated till an adequate amount of periosteum is exposed.
5. A horizontal incision will then be given at the apical extent of the periosteum where it is still attached to the bone.
6. The periosteum will then be separated from the underlying bone and reflected coronally to an extent where it is still attached to the bone.
7. The reflected periosteum will then be inverted such that the cambium layer covers the denuded root.
8. Once the periosteum is in place, it is sutured and secured.
9. The reflected partial thickness flap will be coronally advanced such that it covers the periosteum and will be sutured using a sling suture.
10. The vertical incision will be sutured using an interrupted suture. 8

For group B (control group):

Coronally advanced flap with subepithelial connective tissue graft will be carried out; an envelope flap design will be used according to Zucchelli & De Sanctis 2000 as follows:

1. An intrasulcular incision will be performed involving at least one tooth mesial and at least one tooth distal to the teeth with gingival recessions.
2. Oblique incisions will be traced at the interdental soft tissue level to achieve a coronal rotation of the surgical papilla.
3. The flap will be then raised up to the mucogingival junction (MGJ) with a periosteal elevator and mobilized with a sharp horizontal periosteal incision beyond the MGJ.
4. Exposed root surfaces will be carefully treated with gentle root planing.
5. The anatomic interdental papillae will be carefully de-epithelialized.
6. The split-full-split thickness flap will be then passively positioned above the CEJ of the involved teeth and interrupted or sling sutures were positioned to achieve optimal buccal flap adaptation.
7. The connective tissue graft will be harvested from the palate using the trap door technique (Langer & Langer 1985), adapted to cover each exposed root about 1 mm beyond the CEJ, and stabilized with resorbable sutures.
8. The flap will be then coronally sutured using sling or interrupted sutures.

Post-surgical protocol (Pini-Prato et al.,2010 and Cairo et al., 2016) :

Participants for both groups will be instructed to:

1. Intermittently apply an ice bag for the first 4 hours.
2. Take ibuprofen 600 mg at the end of the surgical procedure and will be instructed to take another tablet 6 h later and additional doses if needed.
3. Avoid any mechanical trauma and tooth-brushing for 3 weeks in the surgical area.
4. Smokers will be reminded to quit smoking during the trial time (6 months).
5. Chlorexidine rinses will be prescribed twice daily for 1 min. seven days after the surgery.
6. Sutures will be removed and prophylaxis will be performed. 9
7. About 3 weeks after surgery, patients will be instructed to resume mechanical tooth-cleaning.

Follow up strategy:

Patients will be recalled after 3and 6 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Gender: Male and Female
2. Age: >20 years
3. Have RT1 and RT2 gingival recession

Exclusion Criteria:

1. Medically compromised
2. History of certain medications
3. Pregnant females
4. Periapical involvement in selected teeth
5. History of periodontal surgery involving experimental teeth
6. If the problem was due to orthodontic treatment

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-01-25 (Estimated); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-08-28 (Estimated)

PRIMARY OUTCOMES:
Post-operative discomfort | 3 weeks
  Numerical using Visual analogue scale (VAS) Questionnaire

SECONDARY OUTCOMES:
Amount of root coverage | 3 months and 6 months
  continuous (mm)
Probing depth | 3 months and 6 months
  continuous (mm)
esthetics | 6 months
  numerical using Root coverage esthetic score (RES)
patient's satisfaction | 6 months
  categorical via assessment of patient-related criteria using a 3-point rating scale

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Faclty of dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
publishing in an international journal
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year